CLINICAL TRIAL: NCT02777593
Title: Evaluation of the GORE® TAG® Thoracic Branch Endoprosthesis (TBE Device) in the Treatment of Lesions of the Aortic Arch and Descending Thoracic Aorta, Zone 2
Brief Title: Evaluation of the GORE® TBE Device in the Treatment of Lesions of the Aortic Arch and Descending Thoracic Aorta, Zone 2
Acronym: SSB 11-02
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSB 11-02 Pivotal (Zone 2)
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Results first posted 2022-11-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Aortic Aneurysm, Thoracic; Aorta; Lesion
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zone 2 Aneurysm (Other): Includes primary (hypothesis-driven) aneurysm cohort and continued access. Subjects enrolled for treatment with the TBE device with proximal implantation in aortic Zone 2.
  Interventions: Device: GORE® TAG® Thoracic Branch Endoprosthesis
- Zone 2 Non-aneurysm (Other): Includes dissection, traumatic transection and other isolated aortic lesion cohorts. Subjects enrolled for treatment with the TBE device with proximal implantation in aortic Zone 2.
  Interventions: Device: GORE® TAG® Thoracic Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® TAG® Thoracic Branch Endoprosthesis — Endovascular repair with the TBE Device

SUMMARY:
The objective of this study is to determine whether the GORE® TAG® Thoracic Branch Endoprosthesis is safe and effective in treating lesions of the aortic arch and descending thoracic aorta, requiring Zone 2 proximal implantation of the device.

DETAILED DESCRIPTION:
For Zone 2, there are two arms (Aneurysm arm, Non-aneurysm arm) and four cohorts, described as follows: Zone 2 Aneurysm, Zone 2 Dissection, Zone 2 Traumatic Transection, and Zone 2 Other Isolated Lesion. Continued access Subjects were enrolled in the Zone 2 Aneurysm arm. The Zone 2 Aneurysm cohort was the only cohort analyzed with a hypothesis test, however data was collected similarly for all cohorts and for continued access Subjects. Zone 2 Subjects enrolled for analysis were from the United States only.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of thoracic aortic pathology deemed to warrant surgical repair which requires proximal graft placement in Zone 0-2.
2. Age ≥18 years at time of informed consent signature
3. Subject is capable of complying with protocol requirements, including follow-up
4. Informed Consent Form (ICF) is signed by Subject or legal representative
5. Must have appropriate proximal aortic landing zone.
6. Must have appropriate target branch vessel landing zone
7. For patients with aneurysm/isolated lesion, must have appropriate distal aortic landing zone.

Exclusion Criteria:

1. Concomitant disease of the ascending aorta or aneurysm of the abdominal aorta requiring repair
2. Previous endovascular repair of the ascending aorta
3. Previous endovascular repair of the DTA with a non-Gore device
4. Surgery within 30 days prior to enrollment, with the exception of surgery for Ascending Aortic Dissection and/or placement of vascular conduit for access
5. Infected aorta
6. Life expectancy <2 years
7. Myocardial infarction within 6 weeks prior to treatment
8. Stroke within 6 weeks prior to treatment, stroke defined as rapidly developing clinical signs of focal (or global) disturbance of cerebral function, lasting more than 24 hours or leading to death, with no apparent cause other than that of vascular origin.
9. Patient has a systemic infection and may be at increased risk of endovascular graft infection
10. Pregnant female at time of informed consent signature
11. Degenerative connective tissue disease, e.g. Marfan's or Ehler-Danlos Syndrome
12. Participation in another drug or medical device study within one year of study enrollment
13. Known history of drug abuse within one year of treatment
14. Presence of protruding and/or irregular thrombus and/or atheroma in the aortic arch or ascending aorta
15. Tortuous or stenotic iliac and/or femoral arteries preventing introducer sheath insertion and the inability to use a conduit for vascular access
16. Planned coverage of celiac artery
17. Patient has known sensitivities or allergies to the device materials
18. Patient has known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment
19. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin
20. Patient with a history of a hypercoagulability disorder and/or hypercoagulability state
21. Diameter taper outside of the device sizing range between proximal and distal landing zones of aorta and the inability to use additional devices of different diameters to compensate for the taper
22. Mycotic aneurysm
23. Persistent refractory shock (systolic blood pressure <90 mm Hg)
24. Patient has body habitus or other medical condition which prevents adequate visualization of the aorta
25. Renal failure defined as patients with an estimated Glomerular Filtration Rate (eGFR) <30 or currently requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Dake, MD, Principal Investigator — Stanford University; Himanshu Patel, MD, Principal Investigator — University of Michigan
Locations (35):
- United States (35):
  - Keck Medical Center of USC, Los Angeles, California
  - Cedar-Sinai Medical Center, Los Angeles, California
  - Leland Stanford Junior University, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - University of Florida - Gainesville, Gainesville, Florida
  - Univeristy of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University of Louisville Jewish Hospital, Louisville, Kentucky
  - University or Maryland Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Research Foundation SUNY Buffalo, Buffalo, New York
  - Carolinas HealthCare Systems, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Cardiovascular Surgery Clinic, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Baylor College of Medicine - Houston, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann, Houston, Texas
  - Heart Hospital at Baylor Plano, Plano, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin System, Madison, Wisconsin

REFERENCES:
- [Derived] Squiers JJ, DiMaio JM, Schaffer JM, Baxter RD, Gable CE, Shinn KV, Harrington K, Moore DO, Shutze WP, Brinkman WT, Gable DR. Surgical debranching versus branched endografting in zone 2 thoracic endovascular aortic repair. J Vasc Surg. 2022 Jun;75(6):1829-1836.e3. doi: 10.1016/j.jvs.2021.12.068. Epub 2022 Jan 5. PMID 34998942

RESULTS

PARTICIPANT FLOW:
Groups:
- Zone 2 Aneurysm Cohort: Aneurysm arm, hypothesis-driven cohort
- Zone 2 Dissection Cohort: Non-aneurysm arm, dissection cohort
- Zone 2 Traumatic Transection Cohort: Non-aneurysm arm, traumatic transection cohort
- Zone 2 Other Isolated Lesion Cohort: Non-aneurysm arm, other isolated lesion cohort
- Zone 2 Aneurysm Continued Access: Aneurysm arm, continued access subjects
Period: Overall Study
Arm/Group | Zone 2 Aneurysm Cohort | Zone 2 Dissection Cohort | Zone 2 Traumatic Transection Cohort | Zone 2 Other Isolated Lesion Cohort | Zone 2 Aneurysm Continued Access
Started | 85 (One participant (who died and is included in the death count within this section) is excluded from results analysis as pre-specified due to a major I/E violation (i.e. drug abuse), n=84 for analysis.) | 136 | 10 (One participant excluded from results analysis as pre-specified (i.e. per FDA request for enrollment into the wrong cohort), n=9 for analysis.) | 13 | 6
Completed | 44 | 54 | 1 | 1 | 0
Not Completed | 41 | 82 | 9 | 12 | 6
Not completed — Still in study | 1 | 32 | 3 | 6 | 5
Not completed — Death | 21 | 28 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 1 | 1 | 0
Not completed — Lost to Follow-up | 8 | 16 | 5 | 0 | 1
Not completed — Physician Decision | 2 | 2 | 0 | 0 | 0
Not completed — Discontinued due to Other | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two participants (1 Zone 2 Aneurysm and 1 Zone 2 Traumatic Transection) that are counted in the Participant Flow section above are excluded from this analysis, as pre-specified, due to a major I/E violation or an FDA-mandated exclusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zone 2 Aneurysm Cohort | Zone 2 Dissection Cohort | Zone 2 Traumatic Transection Cohort | Zone 2 Other Isolated Lesion Cohort | Zone 2 Aneurysm Continued Access | Total
Number analyzed (Participants) | 84 | 136 | 9 | 13 | 6 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (11.1) | 62.7 (11.2) | 42.4 (19.0) | 64.8 (13.3) | 59.8 (15.9) | 64.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 1 | 7 | 3 | 75
  Male | 53 | 103 | 8 | 6 | 3 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 4 | 3 | 0 | 16
  Not Hispanic or Latino | 82 | 127 | 5 | 10 | 6 | 230
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 67 | 99 | 5 | 9 | 5 | 185
  Black or African American | 12 | 29 | 0 | 2 | 1 | 44
  Asian | 3 | 3 | 0 | 0 | 0 | 6
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Hawaiian or Pacific Islander | 1 | 1 | 0 | 0 | 0 | 2
  Other | 1 | 3 | 4 | 2 | 0 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/(m^2)] | 28.8 (6.3) | 30.6 (6.5) | 29.5 (5.0) | 25.8 (5.3) | 36.3 (8.3) | 29.8 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Primary Endpoint Success for Zone 2
Description: Primary Endpoint was composite of the following events: device technical success and absence of aortic rupture, lesion-related mortality, disabling stroke, permanent paraplegia, permanent paraparesis, new onset renal failure requiring permanent dialysis, additional unanticipated post-procedural surgical or interventional procedure related to the device/procedure/withdrawal of the delivery system. Limited to 30 days: disabling stroke, permanent paraplegia, permanent paraparesis, new onset renal failure requiring permanent dialysis.
Time Frame: 12 Months
Population: Two participants (1 Zone 2 Aneurysm and 1 Zone 2 Traumatic Transection) that are counted in the Participant Flow section above are excluded from this analysis, as pre-specified, due to a major I/E violation or an FDA-mandated exclusion.
  Primary Endpoint composite denominator was restricted to number of participants either with a primary endpoint event or imaging performed in the 12 Month window.
Measure: Number; unit: proportion of participants
Arm/Group | Zone 2 Aneurysm Cohort | Zone 2 Dissection Cohort | Zone 2 Traumatic Transection Cohort | Zone 2 Other Isolated Lesion Cohort | Zone 2 Aneurysm Continued Access
Number analyzed (Participants) | 74 | 109 | 6 | 8 | 6
proportion of participants | 0.838 | 0.881 | 1.0 | 0.875 | 1.0
Statistical Analysis 1: Comparison: Zone 2 Aneurysm Cohort; Primary endpoint success was defined as the proportion of analysis-eligible participants without a primary endpoint event and with 12-Month imaging performed. Results were tested against a performance goal (PG) of 0.64 (i.e. 64%), derived from historical GORE TAG® and Conformable TAG® data. Additionally, using a one-sided alpha of 0.05 and Exact Test, minimum power of 80%, the sample needed was 70 patients. With attrition, 85 patients were required; Test type: Other — Performance goal tested using Exact method calculation to estimate the 95% one-sided lower confidence level (95% LCL) on the proportion of participants with primary endpoint success. If the 95% LCL exceeded 0.64, then the the null hypothesis was to be rejected and the PG was met; 95% Exact Lower Confidence Limit = 0.751

ADVERSE EVENTS:
Time Frame: Adverse events collected for 60 Months, rates shown are through all reported follow-up, follow-up is ongoing for participants who have not completed the study.
Description: The two excluded participants (1 Zone 2 Aneurysm and 1 Zone 2 Traumatic Transection due to a major I/E violation or an FDA-mandated exclusion) have been included in this Adverse Events section.
  Collection starting at endovascular procedure
Arm/Group | Zone 2 Aneurysm Cohort | Zone 2 Dissection Cohort | Zone 2 Traumatic Transection Cohort | Zone 2 Other Isolated Lesion Cohort | Zone 2 Aneurysm Continued Access
All-Cause Mortality (participants affected / at risk) | 21/85 | 28/136 | 0/10 | 5/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 61/85 | 99/136 | 3/10 | 9/13 | 4/6
Other Adverse Events (participants affected / at risk) | 74/85 | 111/136 | 7/10 | 11/13 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zone 2 Aneurysm Cohort (N=85) | Zone 2 Dissection Cohort (N=136) | Zone 2 Traumatic Transection Cohort (N=10) | Zone 2 Other Isolated Lesion Cohort (N=13) | Zone 2 Aneurysm Continued Access (N=6)
Acute anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute blood loss anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Anemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemotherapy induced neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemolytic anemia drug-induced (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normocytic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Symptomatic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vaso-occlusive crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction type 2 (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute on chronic heart failure (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aortic valve insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asystole (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation aggravated (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 7 (9) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure aggravated (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic aggravated (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic diastolic heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complete heart block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Heart block AV (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral regurgitation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Persistent atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type II second degree atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unstable angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sickle-cell beta thalassemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Adrenal mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primary hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (left) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataracts (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Detached retina (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiretinal membrane (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden visual loss (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision loss (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Celiac artery aneurysm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Celiac artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohns disease aggravated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum of esophagus, acquired (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ischemic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mesenteric ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurogenic bowel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter related thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (non-cardiac) (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Continued perfusion of a false lumen (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Debility (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Distal aorta false lumen perfusion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Distal branch false lumen perfusion (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Edema lower limb (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Fever of unknown origin (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Slight fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stent thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak type IA (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak type IB (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak type IC (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak type II (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak type III (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unilateral leg swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unknown cause of death (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Unspecified chest pain (General disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular stent-graft occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute exacerbation of chronic bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of leg (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Community acquired pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemophilus parainfluenzae infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Healthcare associated pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal abscess (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Klebsiella pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella septicemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Methicillin-resistant Staphylococcus aureus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Methicillin-resistant Staphylococcus aureus sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericolic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 5 (6) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Spinal osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus aureus bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 6 (9) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vascular graft infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular stent graft infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Broken leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Closed fracture of unspecified part of tibia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device placement at incorrect location (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture of intertrochanteric section of femur, closed (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fractured hip (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured ribs (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Great toe fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemodilution (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural hematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post spinal headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postimplantation syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rupture spleen (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Third degree burns (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cells in cerebrospinal fluid (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia aggravated (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia aggravated (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Protein-calorie malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type II diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volume overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest wall hematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Degenerative spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interscapular pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Olecranon bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in thigh (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff tear arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ductal carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hormone-refractory prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of sigmoid colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvar cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute toxic metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anoxic brain damage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anterior spinal artery syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Carotid artery insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral small vessel ischemic disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Convulsive status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy acute (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracerebral hematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraparenchymal cerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraventricular hemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Near syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nonconvulsive status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Numbness in hand (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paralysis leg (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stroke syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncopal attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Tonic-clonic seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device dislodgement (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device lead fracture (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intensive care unit delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 6 (7) | 0 (0) | 1 (2) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease stage 3 (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney atrophic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney stones (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure aggravated (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal hematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stone urinary bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureter obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteral calculus (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral stricture (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic floor dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deviated nasal septum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flash pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercapnic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hypercarbia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decubitus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pressure ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal aortic aneurysm enlargement (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute limb ischemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aneurysm enlargement (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm enlargement (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection rupture (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aortic intramural hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascending aortic dissection (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Atherosclerotic cardiovascular disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis leg (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep venous thrombosis arm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dissecting aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hemodynamic instability (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhagic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Hypertension worsened (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Iliac artery aneurysm enlargement (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iliac artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliac artery rupture (Vascular disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Iliofemoral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inferior vena cava stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Popliteal artery aneurysm (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Retrograde aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock, unspecified (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic aortic aneurysm (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thoracic aortic aneurysm enlargement (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracoabdominal aortic aneurysm (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thoracoabdominal aortic aneurysm enlargement (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Thromboembolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type A aortic dissection (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Type B aortic dissection (Vascular disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Uncontrolled hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous stasis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zone 2 Aneurysm Cohort (N=85) | Zone 2 Dissection Cohort (N=136) | Zone 2 Traumatic Transection Cohort (N=10) | Zone 2 Other Isolated Lesion Cohort (N=13) | Zone 2 Aneurysm Continued Access (N=6)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Blood loss anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercoagulability (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Long QT syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Tricuspid regurgitation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurry vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Acid reflux (esophageal) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (2) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiatal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mesenteric edema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal hematoma (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial stent occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema of lower extremities (General disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Low grade fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 9 (10) | 8 (10) | 2 (2) | 5 (5) | 0 (0)
Stent-graft endoleak type IA (General disorders) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak type II (General disorders) | 10 (11) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Substernal pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Unilateral leg swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular stent-graft thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weakness generalized (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of leg (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 7 (8) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative pain (Injury, poisoning and procedural complications) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tick bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appetite lost (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Volume overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8) | 0 (0) | 1 (1) | 0 (0)
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy acute (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Numbness in feet (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Numbness in fingers (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Numbness in leg (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Numbness of upper arm (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Numbness of upper extremities (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paresthesia lower limb (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tingling of extremity (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Acute tubular necrosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease stage 3 (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal infarction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteral calculus (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 6 (6) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exercise dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 0 (0) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary collapse (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 0 (0) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ascending aortic aneurysm enlargement (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (6) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 6 (8) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Hypotension symptomatic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iliac artery dissection (Vascular disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Penetrating atherosclerotic ulcer (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT02777593/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT02777593/SAP_003.pdf